CLINICAL TRIAL: NCT01818414
Title: Dilapan-S With Adjunctive Misoprostol for Same-day Second Trimester Dilation and Evacuation: A Randomized Trial
Brief Title: Same-day Dilapan-S With Adjunctive Misoprostol
Acronym: DAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Concerns for safety
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Christy Boraas, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFPRF-112778
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Therapeutic Abortion
Keywords: Misoprostol administration & dosage; Abortion techniques; Abortion Induced methods; Dilatation and Curettage
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Misoprostol; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol (Experimental): Misoprostol 400 mcg buccal 3 hours prior to D&E as an adjunct to same-day Dilapan-S.
  Interventions: Drug: Misoprostol
- Folic Acid (Placebo Comparator): Folic acid 4 mg buccally 3 hours prior to D&E as an adjunct to same-day Dilapan-S
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: Misoprostol — 400 mcg of buccal misoprostol, 3 hours prior to planned D&E
  Other Names: Cytotec
  Arms: Misoprostol
Drug: Folic Acid — 4 mg of buccal folic acid, 3 hours prior to planned D&E
  Other Names: folate, vitamin M, vitamin B9
  Arms: Folic Acid

SUMMARY:
Cervical preparation before second trimester dilation and evacuation (D&E) reduces risks and complications. Osmotic cervical dilators as well as prostaglandin analogues have been studied for cervical preparation. However, the optimal method for cervical preparation, especially for D&E procedures that occur on the same day as cervical preparation, is not known. This study will investigate misoprostol versus placebo as an adjunct to Dilapan-S for cervical preparation for same-day D&E between 16+0 and 20+6 weeks gestation.

HYPOTHESIS: Administration of 400 µg buccal misoprostol compared to placebo at least 3 hours prior to D&E as an adjunct to cervical preparation with Dilapan-S will decrease operative time for same-day D&E performed between 16+0 and 20+6 weeks.

DETAILED DESCRIPTION:
Dilation and evacuation (D&E) is commonly performed for second trimester abortions and management of second trimester intrauterine fetal demise (IUFD). Cervical preparation prior to second trimester D&E increases safety.

Osmotic cervical dilators and prostaglandin analogs are used widely for cervical preparation before second trimester D&E. Osmotic dilators are placed into the cervical canal, radially expand as they absorb moisture and decrease the risk of cervical injury during D&E. Laminaria tents are the most commonly used osmotic dilator for D&E cervical preparation but require N18 h to reach maximum diameter. Dilapan-S®, a synthetic osmotic cervical dilator, has a significant dilation effect 2 h after placement with the majority of expansion occurring in 4-6 h according to the manufacturer.

Misoprostol is the most commonly used pharmacologic cervical preparation for D&E with duration of action between 2 and 4 h after administration. Multiple studies demonstrate the safety of misoprostol before early second trimester abortion. One prospective and four retrospective studies suggest that same-day cervical preparation with Dilapan-S and/or misoprostol for second trimester D&E through 20 weeks is safe and effective. Misoprostol may be less effective when used alone compared to overnight osmotic dilators for cervical preparation later in the second trimester but has adjunctive benefit on cervical dilation and procedure time when used with overnight osmotic dilators between 16 and 24 weeks. The effect appears most pronounced at N19 weeks gestation. No prospective studies have been published examining misoprostol as an adjunct to osmotic dilators for cervical preparation for same-day D&E.

Administration of adjunctive misoprostol with Dilapan-S has the potential to effectively prepare the cervix and decrease operative time for same-day D&E. We compared cervical preparation with Dilapan-S with and without adjunctive buccal misoprostol for same-day D&E between 16 0/7 and 20 6/7 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years (no upper age limit)
* Gestational age between 16+0 and 20+6 weeks gestation on day of D&E with confirmation of gestational age by ultrasound
* Desires D&E for termination of pregnancy or for fetal demise
* Able to provide written informed consent
* Able to comply with study procedures
* English-speaking

Exclusion Criteria:

* Known allergy or contraindication to misoprostol
* Pregnancy with a multiple gestation
* Known bleeding disorder or current anticoagulation therapy (within one month of procedure)
* Active bleeding or hemodynamically unstable at enrollment
* Signs of chorioamnionitis or clinical infection at enrollment
* Signs of spontaneous labor or cervical insufficiency at enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD MPH, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Planned Parenthood of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Univeristy of Pittsburgh, Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edelman AB, Buckmaster JG, Goetsch MF, Nichols MD, Jensen JT. Cervical preparation using laminaria with adjunctive buccal misoprostol before second-trimester dilation and evacuation procedures: a randomized clinical trial. Am J Obstet Gynecol. 2006 Feb;194(2):425-30. doi: 10.1016/j.ajog.2005.08.016. PMID 16458640
- [Background] Goldberg AB, Drey EA, Whitaker AK, Kang MS, Meckstroth KR, Darney PD. Misoprostol compared with laminaria before early second-trimester surgical abortion: a randomized trial. Obstet Gynecol. 2005 Aug;106(2):234-41. doi: 10.1097/01.AOG.0000168629.17326.00. PMID 16055570
- [Background] Newmann SJ, Dalve-Endres A, Diedrich JT, Steinauer JE, Meckstroth K, Drey EA. Cervical preparation for second trimester dilation and evacuation. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD007310. doi: 10.1002/14651858.CD007310.pub2. PMID 20687085
- [Background] Fox MC, Hayes JL; Society of Family Planning. Cervical preparation for second-trimester surgical abortion prior to 20 weeks of gestation. Contraception. 2007 Dec;76(6):486-95. doi: 10.1016/j.contraception.2007.09.004. Epub 2007 Nov 9. PMID 18061709
- [Background] Wilson LC, Meyn LA, Creinin MD. Cervical preparation for surgical abortion between 12 and 18 weeks of gestation using vaginal misoprostol and Dilapan-S. Contraception. 2011 Jun;83(6):511-6. doi: 10.1016/j.contraception.2010.10.004. Epub 2010 Dec 3. PMID 21570547
- [Background] Patel A, Talmont E, Morfesis J, Pelta M, Gatter M, Momtaz MR, Piotrowski H, Cullins V; Planned Parenthood Federation of America Buccal Misoprostol Waiver Group. Adequacy and safety of buccal misoprostol for cervical preparation prior to termination of second-trimester pregnancy. Contraception. 2006 Apr;73(4):420-30. doi: 10.1016/j.contraception.2005.10.004. Epub 2006 Jan 23. PMID 16531179
- [Result] Boraas CM, Achilles SL, Cremer ML, Chappell CA, Lim SE, Chen BA. Synthetic osmotic dilators with adjunctive misoprostol for same-day dilation and evacuation: a randomized controlled trial. Contraception. 2016 Nov;94(5):467-472. doi: 10.1016/j.contraception.2016.05.008. Epub 2016 May 27. PMID 27241895

RESULTS

PARTICIPANT FLOW:
Groups:
- Misoprostol: Misoprostol 400 mcg buccal 3 hours prior to D&E as an adjunct to same-day Dilapan-S.
  Misoprostol
- Folic Acid: Folic acid 4 mg buccally 3 hours prior to D&E as an adjunct to same-day Dilapan-S
  Folic Acid
Period: Overall Study
Arm/Group | Misoprostol | Folic Acid
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misoprostol | Folic Acid | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Operative Time
Description: The primary outcome will be operative time. Operative time will be measured from initial passage of an instrument into the uterus to start the D&E. The end of operative time will be measured by the removal of the last instrument from the uterus to complete the D&E.
Time Frame: Day 1 of the study
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Misoprostol | Folic Acid
Number analyzed (Participants) | 14 | 15
minutes | 11.1 (5.4) | 13.5 (4.0)
Statistical Analysis 1: Comparison: Misoprostol vs Folic Acid; Test type: Superiority or Other; p = 0.17, t-test, 2 sided

2. Secondary Outcome: Patient Pain
Description: Change in pain from baseline to immediately preoperatively using a 100-mm Visual Analogue Scale ("100-mm Visual Analogue Scale with 0 indicating "no pain" and 100 indicating "worst pain in my life")
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Misoprostol | Folic Acid
Number analyzed (Participants) | 14 | 15
mm | 43.9 (25.4) | 24.3 (26.4)
Statistical Analysis 1: Comparison: Misoprostol vs Folic Acid; Test type: Superiority or Other; p = 0.052, t-test, 2 sided

3. Secondary Outcome: Number of Participants With Postoperative Satisfaction
Description: Patient postoperative satisfaction with cervical preparation method
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Misoprostol | Folic Acid
Number analyzed (Participants) | 14 | 15
participants | 10 | 14

4. Secondary Outcome: Number of Providers With Overall Satisfaction
Description: Provider overall satisfaction with cervical preparation
Time Frame: Day 1
Measure: Number; unit: providers
Arm/Group | Misoprostol | Folic Acid
Number analyzed (Participants) | 14 | 15
providers | 10 | 9

5. Secondary Outcome: Complications
Description: Incidence of surgical complications related to D&E
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Misoprostol | Folic Acid
Number analyzed (Participants) | 14 | 15
participants | 0 | 2

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Placebo Comparator: Folic Acid: Folic acid 4 mg buccally 3 hours prior to D&E as an adjunct to same-day Dilapan-S
Arm/Group | Misoprostol | Placebo Comparator: Folic Acid
Serious Adverse Events (participants affected / at risk) | 0/14 | 2/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Misoprostol (N=14) | Placebo Comparator: Folic Acid (N=15)
Hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Cervical laceration during dilation and evacuation procedure resulting in hemorrhage treated with uterine artery embolization
Hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Cervical laceration during dilation and evacuation procedure resulting in hemorrhage treated with hysterectomy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes